CLINICAL TRIAL: NCT07114146
Title: Changes in Heart Rate Variability, Heart Rate, Blood Pressure, and Mood After Walking in Green Spaces. A Comparison of Environments With Healthy Adults.
Brief Title: Physiological and Mood Changes After Walking in Green Spaces. A Comparison of Environments.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vigo (Other)
Responsible Party: Principal Investigator, Ana Gil Iglesias, Principal investigator, Universidade de Vigo
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: ETICA-ULE-087-2025
Record Dates: First submitted 2025-07-28; First posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Healthy Subjects (HS); Forest Therapy; Autonomic Nervous System Activity; Mood
Keywords: Forest therapy; Autonomic nervous system; Mood; forest

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Masking Description: The persons in charge of data extraction and statistics will be masked. The persons in charge of the measurements will also be masked before the transfer of the subjects and after the return of the subjects to the place of departure on the days of exposure; they will not know which exposure each subject will perform on each day of intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- EXPOSURE IN SEQUENCE OF A-B-C-D ENVIRONMENTS (Experimental)
  Interventions: Other: WALK THROUGH ENVIRONMENT A; Other: WALK THROUGH ENVIRONMENT B; Other: WALK THROUGH ENVIRONMENT C; Other: WALK THROUGH ENVIRONMENT D
- EXPOSURE IN SEQUENCE OF B-C-A-D ENVIRONMENTS (Experimental)
  Interventions: Other: WALK THROUGH ENVIRONMENT A; Other: WALK THROUGH ENVIRONMENT B; Other: WALK THROUGH ENVIRONMENT C; Other: WALK THROUGH ENVIRONMENT D
- EXPOSURE IN SEQUENCE OF C-A-B-D ENVIRONMENTS (Experimental)
  Interventions: Other: WALK THROUGH ENVIRONMENT A; Other: WALK THROUGH ENVIRONMENT B; Other: WALK THROUGH ENVIRONMENT C; Other: WALK THROUGH ENVIRONMENT D

INTERVENTIONS:
Other: WALK THROUGH ENVIRONMENT A — A 3 km solo hike at a leisurely walking pace on a path that is easy to walk and has very little elevation gain. Located in Pontevedra Province.
Other: WALK THROUGH ENVIRONMENT B — A 3 km solo hike at a leisurely pace on an easy walking trail with very little elevation gain. Located in the province of Pontevedra.
Other: WALK THROUGH ENVIRONMENT C — 3 km solo hike at a leisurely pace on an easy trail with little elevation gain. Located in the province of Pontevedra.
Other: WALK THROUGH ENVIRONMENT D — Individual 3 km treadmill walk in a closed room facing a wall without pictures or windows at a leisurely walking pace with no gradient. This room will be located on the Pontevedra University Campus.

SUMMARY:
Natural environments, and more specifically forest environments, have shown in the last decade a growing interest as a protection against the frenetic pace of life of a large part of the urban population in developed countries, where symptoms related to stress and anxiety are associated with an increasingly frequent state of sub-health.

The investigators propose to perform a randomized crossover study to analyze the effects of a walk in the forest on physiological and psychological markers related to autonomic nervous system activity in healthy adult. In addition, the investigators intend to observe whether the characteristics and perceptions of the forest environment could affect the results obtained in these markers using a scale created for this purpose.

Participants will be healthy adults with no history of serious physical or psychological illnesses, who will be exposed to three forest environments.

Physiological markers will be measured, including heart rate variability, which will be measured with a heart rate sensor that will monitor data throughout the exposure period, and heart rate and systolic and diastolic blood pressure, which will be measured with an automated device before and after each exposure. Before and after the walk through each of the forest environments, mood will be measured using the POMS scale, and our scale will be used to measure the perceived environmental quality after exposure to each environment.

In addition to the walk through the three forest environments, a control environment on an indoor treadmill will be used as a comparator, where distance, slope and walking speed will be adjusted to replicate the intensity and physical demand of the three outdoor routes.

The four interventions will be organized to create three different exposure sequences. Each exposure sequence will be randomly assigned to a different group. In turn, each participant will be randomly assigned to one of the three groups, so that all participants will undergo all four interventions in a repeated measures design.

Our hypothesis supports the idea that exposure to forest environments causes changes in physiological parameters and mood associated with positive regulation for health and for the autonomic nervous system in healthy adults compared to a neutral non-forest environment. As a second hypothesis, environmental characteristics as well as the perceived quality of the forest environment would be related to the magnitude of such changes associated with autonomic nervous system regulation and mood in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

- Those who have the ability and physical strength to walk 3 km in a calm manner without presenting or consciously suffering any type of adverse symptom.

Exclusion Criteria:

* Pregnancy
* History of severe physical or mental illness
* Drug addiction (including narcotic drugs and non-narcotics) habitual.
* High risk of fall
* Severe outdoor allergies

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
CHANGES IN RR INTERVAL DURING FOREST EXPOSURE | This measurement is carried out each of the four days in which the subjects take a walk in each of the four study places. From 5 minutes before the start of the 3 km walk until 5 minutes after the end of the walk.
  We will measure this variable continuously from 5 minutes before the start of each walk to 5 minutes after the end of each walk.
  The RR interval is a parameter related to Heart Rate Variability, its analysis is commonly used to evaluate the functioning of cardiac autonomic regulation.
CHANGES IN Root Mean Square of Successive Difference Root of RR Interval (RMSSD) DURING FOREST EXPOSURE | This measurement is carried out each of the four days in which the subjects take a walk in each of the four study places. From 5 minutes before the start of the 3 km walk until 5 minutes after the end of the walk.
  We will measure this variable continuously from 5 minutes before the start of each walk to 5 minutes after the end of each walk.
  The RMSSD is a parameter related to Heart Rate Variability, its analysis is commonly used to evaluate the functioning of cardiac autonomic regulation.
CHANGES IN standard deviation of RR intervals (SDNN) DURING FOREST EXPOSURE | This measurement is carried out each of the four days in which the subjects take a walk in each of the four study places. From 5 minutes before the start of the 3 km walk until 5 minutes after the end of the walk.
  We will measure this variable continuously from 5 minutes before the start of each walk to 5 minutes after the end of each walk.
  The SDNN is a parameter related to Heart Rate Variability, its analysis is commonly used to evaluate the functioning of cardiac autonomic regulation.
CHANGES IN High frequency component (HF) DURING FOREST EXPOSURE | This measurement is carried out each of the four days in which the subjects take a walk in each of the four study places. From 5 minutes before the start of the 3 km walk until 5 minutes after the end of the walk.
  We will measure this variable continuously from 5 minutes before the start of each walk to 5 minutes after the end of each walk.
  The HF component is a parameter related to Heart Rate Variability, its analysis is commonly used to evaluate the functioning of cardiac autonomic regulation.
CHANGES IN Low frequency component (LF) DURING FOREST EXPOSURE | This measurement is carried out each of the four days in which the subjects take a walk in each of the four study places. From 5 minutes before the start of the 3 km walk until 5 minutes after the end of the walk.
  We will measure this variable continuously from 5 minutes before the start of each walk to 5 minutes after the end of each walk.
  The LF component is a parameter related to Heart Rate Variability, its analysis is commonly used to evaluate the functioning of cardiac autonomic regulation.
CHANGES IN Sympathovagal balance (LF/HF) DURING FOREST EXPOSURE | This measurement is carried out each of the four days in which the subjects take a walk in each of the four study places. From 5 minutes before the start of the 3 km walk until 5 minutes after the end of the walk.
  We will measure this variable continuously from 5 minutes before the start of each walk to 5 minutes after the end of each walk.
  The sympathovagal balance is a parameter related to Heart Rate Variability, its analysis is commonly used to evaluate the functioning of cardiac autonomic regulation.
CHANGES IN HEART RATE | This measurement is carried out each of the four days in which the subjects take a walk in each of the four study places: Baseline (min 0), 5 minutes pre walk, 5 minutes post walk and after the period of time corresponding to the vehicle journey.
  We will measure this variable punctually on four occasions each of the 4 days of intervention. This data will be taken with an Automated Blood Pressure Device placed on the left arm with participants resting in a seated position. Each measurement is taken three times. Participants rest for 5 minutes before the measurements.
CHANGES IN SYSTOLIC BLOOD PRESSURE | This measurement is carried out each of the four days in which the subjects take a walk in each of the four study places: Baseline (min 0), 5 minutes pre walk, 5 minutes post walk and after the period of time corresponding to the vehicle journey.
  We will measure this variable punctually on four occasions each of the 4 days of intervention. This data will be taken with an Automated Blood Pressure Device placed on the left arm with participants resting in a seated position. Each measurement is taken three times. Participants rest for 5 minutes before the measurements.
CHANGES IN DIASTOLIC BLOOD PRESSURE | This measurement is carried out each of the four days in which the subjects take a walk in each of the four study places: Baseline (min 0), 5 minutes pre walk, 5 minutes post walk and after the period of time corresponding to the vehicle journey.
  We will measure this variable punctually on four occasions each of the 4 days of intervention. This data will be taken with an Automated Blood Pressure Device placed on the left arm with participants resting in a seated position. Each measurement is taken three times. Participants rest for 5 minutes before the measurements.
CHANGES IN THE PROFILE OF MOOD STATES. SHORT SPANISH VERSION | This measurement is carried out each of the four days in which the subjects take a walk in each of the four study places: Baseline (min 0) and post walk immediately after finishing physiological measurements
  We will measure this variable punctually on two occasions each of the 4 days of intervention. The POMS is a questionnaire for the measurement of mood. POMS is a reliable and valid psychometric instrument that includes 30 adjectives in this Spanish short versions, rated on a scale of 0-4 (0 = none; 4 = very strong), which can be integrated into six factors, four of these factors are negative: Anger, Fatigue, Tension and Depressed State; and two are positive: Vigour and Friendship.
CHANGES IN TOTAL MOOD DISTURBANCE | This measurement is carried out each of the four days in which the subjects take a walk in each of the four study places: Baseline (min 0) and post walk immediately after finishing physiological measurements
  We will measure this variable punctually on two occasions each of the 4 days of intervention. Total Mood Disturbance TMD It is a score that measures a person's emotional distress, psychological distress or subjective well-being. It can be obtained from POMS results; it is calculated from the sum of all the values obtained for each factor, with the exception of the two positive factors, which are subtracted.
SCALE OF PERCEIVED ENVIRONMENTAL QUALITY OF THE FOREST ENVIRONMENT | This measurement is performed on each of the three days when subjects take a walk in each of the three outdoor study environments: Post walk, immediately after completing the physiological measurements.
  We will measure this variable once each of the 4 days of intervention. We will use the "Scale of perceived environmental quality of the forest environment", a 41-question recording method to determine the quality perceived by the respondent of a given forest environment.
  It is configured by means of a series of questions in which the person quantitatively rates certain characteristics of the tree stands according to his or her own criteria. 39 of the questions use a 5-point Likert scale in which each question is rated from 1 to 5, with 1 = Not at all, and 5 = Very much. Questions 40 and 41 are called criterion questions where on a scale of 1 to 10 the person responds according to his or her criteria 1 = very low/very little and 10 = outstanding.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad de Vigo. Campus Pontevedra, Pontevedra, Pontevedra, Spain

IPD SHARING:
Plan to Share IPD: Undecided